CLINICAL TRIAL: NCT03750500
Title: Clinical Impact of a Digital Home-based Falls Prevention Program on Elderly People - a Randomized Controlled Trial
Brief Title: Clinical Impact of a Digital Home-based Falls Prevention Program on Elderly People
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SH-RCT-FP-01
Record Dates: First submitted 2018-11-20; First posted 2018-11-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Fall
MeSH Terms: interventions — Medication Review

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants included in this arm will benefit from a 12-week exercise program using the novel biofeedback rehabilitation device, under remote monitoring from a physical therapist
  Interventions: Device: Biofeedback device; Behavioral: Education on falls risk; Other: Medication review; Diagnostic Test: Visual and auditory screening
- Standard of Care (Placebo Comparator): Patients included in this arm will benefit from the standard of care currently in place in the Primary Care facility: education on risk factors for falls, medication review, visual and auditory acuity screening.
  Interventions: Behavioral: Education on falls risk; Other: Medication review; Diagnostic Test: Visual and auditory screening

INTERVENTIONS:
Device: Biofeedback device — 12-week exercise program performed through the device
  Other Names: SWORD Phoenix
  Arms: Experimental
Behavioral: Education on falls risk — Education on falls risk factors and how to minimize them
Other: Medication review — Medication will be reviewed to reduce sedative drugs and minimize interactions
Diagnostic Test: Visual and auditory screening — Patients will go through visual and auditory screening as part of their regular care

SUMMARY:
This study is a single-center, prospective, non-blind, parallel-group, randomized controlled trial with an experimental and a control group with the aim of evaluating the clinical impact of a home-based falls prevention program using a new biofeedback system on community-dwellers older adults with fall risk in comparison with standard of care.

The experimental group will perform a 12-week exercise program at home, under remote monitoring from a clinical team, whereas the control group will benefit from standard medical care currently in place at the participating primary care facility.

The hypothesis is that the home-based falls prevention program will lead to a lower risk of falling than standard medical care.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 65 years old
2. Ability to walk at least 20 meters, unaided or with unilateral support
3. Ability to understand motor complex commands
4. Mini-Mental State Examination (MMSE) score > 24 points
5. Functional independence for instrumental activities of daily living
6. Risk of recurrent falls, defined as 5xSST score > 15,00 seconds

Exclusion Criteria:

1. Patients residing in nursing homes, daycare units or assisted-living facilities
2. Aphasia, dementia or psychiatric comorbidity, significantly interfering with communication or compliance with a home-based exercise program
3. Severe visual our hearing, interfering with communication or with compliance to a home-based exercise program
4. Cardiac, respiratory or other condition incompatible with at least 30 minutes of light to moderate physical activity
5. Osteoarticular conditions (e.g. severe osteoarthrosis), which prevent the patient from complying with a home-based exercise program
6. Patients with neurologic conditions (e.g. stroke, multiple sclerosis, Parkinson's disease)
7. Other medical complications, which prevent the patient from complying with a home-based exercise program
8. Illiteracy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in the 5 Times Sit to Stand Test | Baseline; week 4; week 8; week 12 and then week 24
  The 5 Times Sit to Stand Test is a performance test that measures the strength and the lower limb mobility. It consists of the time it takes to stand up from a chair five consecutive times. A cutoff value of 15 seconds is used to distinguish between individuals with and without risk of recurrent falls

SECONDARY OUTCOMES:
Change in the Timed Up and Go Test score | Baseline; week 4; week 8; week 12 and then week 24
  The TUG is a performance test that assesses the mobility, balance and gait in elderly individuals, consisting of the time it takes to stand up from a chair, walk 3 meters, turn around, come back and sit down again.
Change in the Berg Balance Scale | Baseline; week 4; week 8; week 12 and then week 24
  The Berg Balance Scale was developed to evaluate the static and dynamic balance in three domains: sitting, standing and changing posture. It is a scale composed of 14 items graded by an external observer on 5 levels (from 0 to 4). Scale scores range from 0 to 56, with higher scores representing a higher level of functionality.
Change in the Shorts Falls Efficacy Scale-International | Baseline; week 4; week 8; week 12 and then week 24
  The Shorts Falls Efficacy Scale-International was developed in order to systematize on a scale the fear of falling. It is a questionnaire of 7 items filled by the user, evaluating from 1 to 4 the fear of falling during the execution of a series of activities of daily living. It is a standardized and comparable measure over time, which provides an additional dimension in the characterization of participants. The cutoff levels are: low fear (7-8); moderate fear (9-13) and high fear (14-28).

CONTACTS AND LOCATIONS:
Locations (1):
- USF Aldoar, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study aggregate results (including anonymised individual patient data) will be made available
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available upon study publication, for 5 years.
Access Criteria: The protocol will be made available through this platform.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-11-14): https://cdn.clinicaltrials.gov/large-docs/00/NCT03750500/Prot_SAP_ICF_000.pdf